CLINICAL TRIAL: NCT04112966
Title: Manual Lymph Drainage in the Prevention of Lymphedema Related to Breast Cancer
Brief Title: Lymphedema Prevention in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ECA-DLM-5
Record Dates: First submitted 2019-07-22; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer; Lymphedema
Keywords: Lymphedema; Prevention
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Manual Lymph Drainage (Experimental): 14 sessions of manual lymphatic drainage technique in the three months following surgery and received health education on the prevention of lymphedema.
  Interventions: Procedure: 14 sessions of manual lymphatic drainage technique; Other: the health education
- Health education for lymphedema prevention (Other): Only the health education for lymphedema prevention.
  Interventions: Other: the health education

INTERVENTIONS:
Procedure: 14 sessions of manual lymphatic drainage technique — Early manual lymph drainage including 14 sessions of manual lymphatic drainage technique in the three months following surgery and health education for lymphedema prevention including verbal instructions and written materials.
  Arms: Early Manual Lymph Drainage
Other: the health education — The health education for lymphedema prevention.

SUMMARY:
OBJECTIVE: To find out the effectiveness of early application of Manual Lymph Drainage in the prevention of upper limb lymphedema after breast surgery and axillary lymphadenectomy in women with breast cancer.

DESIGN: Randomized, controlled and single blinded clinical trial. Five years duration. Patients were randomly assigned to one of these groups: Experimental group: Manual Lymph Drainage + training in means of prevention; Control group: just training in means of prevention. In both groups several physical therapy assessments were undertaken: 1st before surgery; 2nd 3 month after surgery; 4th, 5th, 6th, 7th, 8th and 9th after 6, 12, 24, 36, 48 and 60 months.

SUBJECTS: Women with breast cancer treated with breast surgery including axillary lymphadenectomy in Provincial Hospital of Toledo, provided that there is no contraindication for manual lymph drainage, and after reading, understanding and freely signing an informed consent form.

SAMPLE SIZE: A total of 150 subjects were included in the study (57 subjects in experimental group and 93 in control group), assuming a 20% of drop-outs and at least 25% reduction, with a statistical power of 75%.

DATA ANALYSIS: To find out the effectiveness of intervention the investigators will compare the rate of lymphedema in both groups by means of a logistic regression analysis, in which the main factor is the intervention group. Other factors aimed to control the effect of the intervention will also be included. In order to compare the rate of appearance of lymphedema in both groups, a survival analysis will also be included.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of breast cancer.
* Undergoing unilateral surgery with axillary lymph-node dissection.

Exclusion Criteria:

* Bilateral breast cancer.
* Systemic disease.
* Locoregional recurrence.
* Any contraindication to physical therapy.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-05 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Circumference measurements | 0 months
  Circumference measurements of the upper limbs using at 5 cm intervals from the elbow fold preoperatively prior to randomization.
Circumference measurements | 3 months
  Circumference measurements of the upper limbs using at 5 cm intervals from the elbow fold preoperatively prior to randomization and then post-operatively on 3 months after surgery.
Circumference measurements | 6 months
  Circumference measurements of the upper limbs using at 5 cm intervals from the elbow fold preoperatively prior to randomization and then post-operatively on 6 months after surgery.
Circumference measurements | 12 months
  Circumference measurements of the upper limbs using at 5 cm intervals from the elbow fold preoperatively prior to randomization and then post-operatively on 12 months after surgery.
Circumference measurements | 24 months
  Circumference measurements of the upper limbs using at 5 cm intervals from the elbow fold preoperatively prior to randomization and then post-operatively on 24 months after surgery.
Circumference measurements | 36 months
  Circumference measurements of the upper limbs using at 5 cm intervals from the elbow fold preoperatively prior to randomization and then post-operatively on 36 months after surgery.
Circumference measurements | 48 months
  Circumference measurements of the upper limbs using at 5 cm intervals from the elbow fold preoperatively prior to randomization and then post-operatively on 48 months after surgery.
Circumference measurements | 60 months
  Circumference measurements of the upper limbs using at 5 cm intervals from the elbow fold preoperatively prior to randomization and then post-operatively on 60 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Romay Barrero, Prof. PhD., Principal Investigator — University of Castilla-La Mancha
Locations (1):
- Provincial Hospital, Toledo, Spain